CLINICAL TRIAL: NCT06410547
Title: Using Large Language Models Such As GPT-4 to Assess Guideline Adherence in Patients with Chronic Obstructive Pulmonary Disease
Acronym: IMPL-AI-MENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Matthias Gröschel, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EA2/322/23
Record Dates: First submitted 2024-04-24; First posted 2024-05-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention (No Intervention): This arm will be treated as usual. No intervention will be performed.
- LLM Assessement (Active Comparator): During hospital stay and after written informed consent, an LLM is asked to indicate if the treatment the patient receives is guideline-concordant. The information is ascertained by two study physicians (human-in-the-loop) and later provided to the treating physician who can recommend a change in therapy to the patient (outside of the study).
  Interventions: Other: LLM

INTERVENTIONS:
Other: LLM — A LLM-based comparison between treatment and guideline.
  Arms: LLM Assessement

SUMMARY:
According to studies in the US and the Netherlands, 33-40% of patients with chronic conditions receive care that does not follow guideline recommendations. These findings have also been demonstrated in the management of COPD. This leads to under- or over-treatment of patients and, in the case of COPD, to exacerbations and hospitalisations. These exacerbations are a significant clinical problem, affecting patient's lung function, quality of life and mortality. They are also a burden on the healthcare system. Technological advances in artificial intelligence offer the opportunity to address these issues in COPD management. In the past year, there have been remarkable innovations in the field of natural language processing, especially through large language models such as GPT-4 from OpenAI and Bard or Gemini from Google. These models offer an opportunity to improve the implementation of evidence-based care in clinical practice.

This study is a prospective, randomised trial that will compare therapy on discharge for patients with COPD. One arm will receive no intervention, while the other arm will receive a treatment recommendation from an LLM. The study will compare the percentage of patients treated according to the guideline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Consent
* Discharge after hospitalization

Exclusion Criteria:

* Lack of Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to treatment guidelines at the time of hospital discharge | From date of admission (which is enrollment) to the date of discharge, assessed up to one month
  The primary endpoint will assess whether the treatment at the time of discharge is consistent with the guidelines' recommendations. This is a binary outcome measure of yes or no.
Percentage of patients treated in concordance with treatment guidelines at the time of hospital discharge | From date of admission (which is enrollment) to the date of discharge, assessed up to one month
  This primary endpoint will assess the percentage of guideline-concordant treatments in each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Gröschel, MD PhD, Principal Investigator — Charité
Locations (1):
- Charité University, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).